CLINICAL TRIAL: NCT02039115
Title: Reduction in Symptomatic Esophageal Stricture Formation Post-two Stage Complete Barrett's Excision for High Grade Dysplasia or Early Adenocarcinoma With Short-term Steroid Therapy: A Randomized, Double-blinded, Placebo-controlled, Multicenter Trial.
Brief Title: Reduction in Symptomatic Esophageal Stricture Formation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closed for low enrollment and the inability to complete the study.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 461672
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Stenosis
MeSH Terms: conditions — Esophageal Stenosis | interventions — Prednisone; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisone (Experimental): Daily oral prednisone is taken for 6 weeks, at a dose of 40mg/day in week 1, 30mg/day in week 2, 20mg/day week 3 and 4, 10mg/day in week 5, and 5mg/day in week 6. Prednisone is taken in the morning. Treatment commences the day of the procedure, with the dose taken with a sip of water prior to discharge. The 6-week treatment regimen is given after both the 1st and 2nd stage complete Barretts excision.
  Interventions: Drug: prednisone
- placebo (Placebo Comparator): Placebo tablets will be taken in the same manner as the prednisone arm.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prednisone — 6 weeks of prednisone and placebo therapy will be given over 6 weeks after both the first and second stage complete Barretts Excision.
  Other Names: steroid
  Arms: prednisone
Drug: placebo — 6 weeks of placebo therapy will be given in the same manner as the prednisone arm after the first and second stage complete Barretts excision.
  Other Names: control
  Arms: placebo

SUMMARY:
Complete endoscopic resection of early neoplastic Barrett's Esophagus (BE) is a curative procedure. However, a significant proportion of patients develop symptomatic esophageal strictures following Complete Barrett's Eradication (CBE), and this limits the technique, particularly for circumferential and longer segment disease. Oral steroid therapy may reduce stricture formation; thereby allowing CBE to be performed with minimal associated morbidity.

DETAILED DESCRIPTION:
The main objective of the proposed randomized trial is to compare the rate of symptomatic oesophageal strictures in patients receiving placebo versus oral prednisone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Barretts mucosa with high grade dysplasia or early esophageal adenocarcinoma (T1a, intramucosal adenocarcinoma).
2. Barretts segment ≥ 30% circumference, ≤C3 and ≤M5.
3. The general health condition of the patient permits anesthesia for endoscopy.
4. Patient is 18 years of age or older.
5. Informed consent is obtained

Exclusion Criteria:

1. Previous (referral) biopsies show low grade dysplasia only, or invasive adenocarcinoma.
2. Barretts segment <30% circumference, >C3 or >M5.
3. During initial gastroscopy there are highly suspicious areas for submucosal invasive cancer (Kudo pit pattern type V; excavated/depressed type morphology; large smooth or ulcerated nodule). In cases of significant doubt, initial resection is of the highly suspicious area only, and urgent histology processing requested. If submucosal invasion is excluded, the patient is rebooked for 1st stage complete barrett's excision (60% circumferential resection) and randomization after a 4-6 weeks interval.
4. Presence of a tight peptic oesophageal stricture that impedes safe and effective endoscopic mucosal resection using a cap (Cook Medical).
5. Active malignancy, uncontrolled Diabetes Mellitus, active or untreated major psychiatric disorder, uncontrolled infection, uncontrolled hypertension, uncontrolled or severe congestive cardiac failure, non-correctable coagulopathy (INR>2, or platelet count <60 x 109/L), osteoporosis, recent peptic ulcer disease, moderate-to-severe glaucoma or untreated glaucoma, or pregnancy.
6. Unable to provide informed consent
7. Allergy to compound used in tablet formulation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hawes Hawes, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prednisone | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stricture Formation
Description: Primary outcome measure is the rate of symptomatic esophageal stricture formation.
Time Frame: 98 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Prednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes